CLINICAL TRIAL: NCT00042796
Title: A Phase I Study Of Decitabine (DAC) (IND # 50733) In Children With Relapsed Or Refractory Acute Leukemia
Brief Title: Decitabine in Treating Children With Relapsed or Refractory Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01873; ADVL0114; U01CA097452 (NIH); CDR0000069471 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Promyelocytic Leukemia (M3); Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Decitabine

ARMS (1):
- Treatment (decitabine) (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 4-6 weeks for a minimum of 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. This phase I trial is studying the side effects and best dose of decitabine in treating children with relapsed or refractory acute myeloid leukemia or acute lymphoblastic leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of decitabine that is associated with consistent evidence of deoxyribonucleic acid (DNA) demethylation in children with relapsed or refractory acute myeloid leukemia or acute lymphoblastic leukemia.

II. Determine the dose-limiting toxicity, pharmacokinetics, and antitumor activity of this drug in these patients.

III. Determine the biologic correlates of decitabine-induced DNA demethylation by characterizing, before and after treatment, global and specific DNA methylation status (using methylation microarrays) and hemoglobin F levels in these patients.

IV. Determine the biologic correlates of decitabine-induced DNA demethylation by characterizing, before and after treatment, global changes in gene expression profiles using cDNA microarrays and drug sensitivity of blast cells by MTT assays in these patients.

V. Determine the biologic correlates of decitabine-induced DNA demethylation by characterizing, before and after treatment, deletions and single nucleotide polymorphisms in genomic DNA of deoxycytidine kinase and cytidine deaminase genes in these patients.

VI. Determine the biologic correlates of decitabine-induced DNA demethylation by characterizing, before and after treatment, acetylation and methylation of histones H3 and H4 and helicase protein expression in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to disease type (acute myeloid leukemia vs acute lymphoblastic leukemia).

Patients receive decitabine IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 4-6 weeks for a minimum of 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 15-21 patients will be accrued for this study within 7.5-21 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed acute myeloid leukemia (AML) or acute lymphoblastic leukemia that is considered refractory to conventional therapy or for which no conventional therapy exists
* For patients with AML:

  * M3 marrow
  * M2 marrow with at least 15% blasts
  * Secondary AML allowed
* CNS involvement allowed
* Performance status - Karnofsky 50-100% (age 17 to 21)
* Performance status - Lansky 50-100% (age 16 and under)
* At least 8 weeks
* See Chemotherapy
* WBC no greater than 30,000/mm^3
* Patients with granulocytopenia, anemia, and/or thrombocytopenia are eligible but are not evaluable for hematological toxicity
* Bilirubin no greater than 1.5 times normal
* ALT no greater than 5 times normal
* Albumin at least 2 g/dL
* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate at least lower limit of normal
* Shortening fraction at least 27% by echocardiogram
* Ejection fraction at least 50% by MUGA scan
* No evidence of dyspnea at rest
* No exercise intolerance
* Oxygen saturation greater than 94% by pulse oximetry
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Concurrent seizure disorder allowed if well controlled on anticonvulsants
* No grade 2 or greater CNS toxicity
* No uncontrolled infection (i.e., infections associated with fever, dissemination, hemodynamic instability [requiring pressor support], and progression while on therapy)
* No active graft-versus-host disease (GVHD)

  * GVHD well controlled on cyclosporine allowed
* Recovered from prior immunotherapy
* At least 1 week since prior biologic agents
* At least 6 months since prior allogeneic bone marrow transplantation (BMT)
* At least 3 months since prior autologous BMT
* No concurrent sargramostim (GM-CSF)
* No concurrent prophylactic filgrastim (G-CSF) during the first course of therapy
* Recovered from prior chemotherapy
* At least 4 weeks since prior cytarabine
* At least 24 hours since prior cytoreductive therapy with hydroxyurea (20-30 mg/kg/day for no more than 7 days) to lower the WBC to no greater than 30,000/mm^3
* No concurrent intrathecal therapy during the first course of decitabine
* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 weeks since prior cranial or craniospinal radiotherapy
* No concurrent medications that induce cytidine deaminase or deoxycytidine kinase (e.g., cytarabine)
* No concurrent medications that mask poor or deteriorating organ function
* No concurrent CNS prophylaxis during the first course of decitabine
* Concurrent anticonvulsants with no known interactions with decitabine allowed
* Concurrent antibacterial or antifungal therapies for controlled infections allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2002-12; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
MTD defined as the highest dose at which fewer than one-third of patients experience DLT assessed using CTC version 2.0 | 4 weeks

SECONDARY OUTCOMES:
CR rate | Up to 3 years
  Will be estimated by proportions.
PR rate | Up to 3 years
  Will be estimated by proportions.
DNA methylation | Up to 3 years
  Pearson correlation will be used.
Gene expression profiles | Up to 3 years
  Will be analyzed using hierarchical clustering.
HDAC/HAT activity | Up to 3 years
  Pearson correlation coefficient analysis will be used.
Presence of mutant helicases | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Norman Lacayo, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States